CLINICAL TRIAL: NCT00004307
Title: Therapeutic and Metabolic Studies of Urea Cycle Disorders: Part A: Nitrogen Flux and Ureagenesis; Part B (Closed): Phase I Adenovirus Vector-Mediated Gene Therapy for Ornithine Transcarbamylase Deficiency
Brief Title: Study of Treatment and Metabolism in Patients With Urea Cycle Disorders
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Baylor College of Medicine (Other)
Purpose: Treatment
Other Study IDs: NCRR-M01RR00188-0606; BCM-H4379
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Amino Acid Metabolism, Inborn Errors
Keywords: inborn errors of metabolism; rare disease; urea cycle disorder
MeSH Terms: conditions — Amino Acid Metabolism, Inborn Errors; Metabolism, Inborn Errors; Rare Diseases; Urea Cycle Disorders, Inborn | interventions — Proteins; Caloric Restriction

INTERVENTIONS:
Behavioral: Protein and calorie controlled diet
Genetic: Ornithine transcarbamylase vector

SUMMARY:
RATIONALE: The urea cycle is the process in which nitrogen is removed from the blood and converted into urea, a waste product found in urine . Urea cycle disorders are inherited disorders caused by the lack of an enzyme that removes ammonia from the bloodstream. Gene therapy is treatment given to change a gene so that it functions normally. Studying the treatment and metabolism of patients with urea cycle disorders may be helpful in developing new treatments for these disorders.

PURPOSE: Two-part clinical trial to study the treatment and metabolism of patients who have urea cycle disorders.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This protocol involves 2 clinical studies. Part A is a metabolic study of glutamine conversion to urea at different levels of protein intake, while on and off medications. Part B is a dose escalation study of a first-generation adenoviral vector with an E1 deletion and an E3 deletion substitution (d1309) expressing ornithine transcarbamylase (OTC).

In Part A, diet is controlled for protein and calories. Intravenous glutamine and urea are administered. Controls are given intravenous arginine, phenylacetate, and benzoate.

In Part B, groups of 3 patients are given a single low, intermediate, or high dose of intravenous OTC vector. Allopurinol is administered every 12 hours for 12 days. As of 12/10/1999, Part B of the study is closed.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

Part A. Patients at least 6 months old with ornithine transcarbamylase deficiency (OTC), i.e.: Hemizygous OTC or homozygous autosomal recessive disorder with evidence of complete enzyme deficiency Hemizygous OTC male with late presentation and presumed evidence for residual enzyme activity OTC heterozygotes (molecular diagnosis) with severely symptomatic to asymptomatic disease Obligate heterozygotes for autosomal recessive disorder (parent or genotyped sibling) Normal adult volunteers and genotyped siblings entered as controls Part B. Metabolically stable heterozygous OTC females aged 18 to under 65 Orotic acid level at least 5 times normal on allopurinol Symptoms ranging from severe to asymptomatic acceptable No prior hospitalization for hyperammonemia Exclusion criteria (Parts A and B): Acute or chronic intercurrent illness Pregnancy Acute hyperammonemia

Ages: 6 Months to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 66
Dates: Start 1999-12

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Lee, Study Chair — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States